CLINICAL TRIAL: NCT05806255
Title: Remote Self-Reporting of Symptoms by Patients With Palliative Care Needs (RELIEF): A Mixed-Methods Implementation Study
Brief Title: Implementation of RELIEF for Patients With Palliative Care Needs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: William Osler Health System (Other)
Collaborators: Humber River Hospital (Other); The Ottawa Hospital (Other); Bruyère Health Research Institute. (Other); University of Ottawa (Other); Ottawa Hospital Research Institute (Other); University of Toronto (Other); Queen's University (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3525
Record Dates: First submitted 2023-03-03; First posted 2023-04-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Palliative Care
Keywords: palliative care; end of life care; e-health tool; implementation science; home care; virtual care; remote monitoring; symptom reporting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RELIEF Intervention Group (Experimental): The RELIEF App will be implemented according to a standardized procedure at the six following sites, with 100 patients recruited at each site:
  1. Home and Community Care Support Services Central West
  2. Home and Community Care Support Services Central
  3. Home and Community Care Support Services Champlain
  4. Home and Community Care Support Services North East
  5. Curve Lake First Nation (CLFN)
  6. St. Mary's Hospital
  Interventions: Device: The RELIEF App

INTERVENTIONS:
Device: The RELIEF App — RELIEF is a virtual app designed for the remote self-reporting of symptoms in patients with palliative care needs. The patient/caregiver securely logs into the site and self-reports symptoms, distress, and pain using the validated clinical tools ESAS-r, Distress Thermometer (DT), and Brief Pain Inventory (BPI) currently in daily use by healthcare providers across Canada.
  This data is reported to the healthcare providers via RELIEF. Any increases in symptom burden, distress, or pain are flagged for clinical review as RELIEF alerts. Healthcare providers received alerts via secure email for any sudden changes in symptom status, or if the patient's symptoms, distress, or pain severity increases by set amounts over a period of time. Following review of the RELIEF alert by the healthcare providers, patients receive (1) earlier intervention; (2) mobilization of auxiliary services; and (3) recommendation for urgent clinic/home visit or emergency department visit.
  Other Names: RELIEF

SUMMARY:
For patients with palliative care needs, access to care is constrained by health system resources and a requirement to visit their clinician for assessments. As assessments typically only occur every 4-8 weeks, this results in emergency department visits by patients/caregivers. More frequent assessments would provide more timely and earlier interventions for patients by their clinicians should intervention be required. However, a key barrier to effective symptom management and patient/family comfort is the lack of real-time symptom status.

RELIEF allows for the remote self-reporting of symptoms by patients to their healthcare providers. It is an easy and effective method of remote symptom reporting for patients with palliative care needs, and RELIEF has the potential to result in significant healthcare cost avoidance and improved patient care. The proposed study will establish the feasibility of implementing RELIEF across a diverse set of populations and settings in Canada.

DETAILED DESCRIPTION:
Over 90% of Canadians agree patients have the right to receive care in their own homes at the end of life and over half of Canadians expect the bulk of their end-of-life care to occur in their own homes. A primary challenge to achieving these outcomes is insufficient resources and services around symptom assessment, monitoring, and management. Poor symptom monitoring in the home and late referrals for symptom management may account for many patients dying in hospitals-nearly 65% of patients in Ontario died in hospitals in 2015/16. Receipt of palliative care services in the home has been associated with a 47% reduction in the likelihood of dying while in hospital. Additionally, costs to the healthcare system are substantially higher in hospitalized patients.

Studies have demonstrated how remote monitoring of symptoms can improve care in patients with palliative care needs. However, some existing digital solutions are limited in that they are rarely well-integrated into the workflow. Additionally, alerting mechanisms to trigger interventions are often absent and the target populations tend to only focus on patients with cancer. Therefore, RELIEF was introduced as an online application designed for the remote self-reporting of symptoms in all patients with palliative care needs. The patient/caregiver securely logs into the site and self-reports symptoms, distress, and pain using validated clinical tools. Results are reported to the patient's healthcare team and flares in symptom burden are flagged for clinical review. These frequent assessments allow for: (1) earlier intervention; (2) mobilization of auxiliary services; and (3) recommendation for emergency or palliative intake. Clinicians and nursing staff access patients' data through RELIEF and receive alerts for any sudden, unexpected, and large changes in symptom status, allowing for timely acute interventions or close passive monitoring, reducing patient stress through the knowledge that their healthcare provider is monitoring their symptoms.

In a small pilot study of RELIEF in just 20 patients, it was found that the patient compliance rate was >80%, with 92% of clinicians reporting improved confidence in the care provided, and an estimated healthcare cost avoidance of over $20,000 per patient over several months was achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has palliative care needs
2. Any life-limiting diagnosis (including non-cancer diagnoses)
3. Score of 40% or above on the Palliative Performance Scale
4. Able to communicate in English or French
5. Have access to the internet
6. Are comfortable learning to use RELIEF for remote symptom self-reporting OR have a caregiver who is comfortable learning to use RELIEF and regularly reporting the patient's symptoms

Exclusion Criteria:

1. Moderate to severe confusion due to delirium or dementia as determined by the patient's healthcare provider
2. A patient with low technology literacy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Daily symptom self-report completed. | Up to 6 months across implementation.
  The percentages of patient who completed questionnaires.
Site adoption. | Immediately after the intervention.
  The number of sites who have implemented RELIEF.
Improved palliative care access. | Immediately after the intervention.
  The percentage of participating patients who actually enrolled in RELIEF study. Descriptive statistics will be used.
Acceptability: Partner sites perceive RELIEF to be agreeable, palatable, and/or satisfactory. | Up to 6 months across implementation.
  CFIR interviews and Hexagon Tool will be used and analyzed qualitatively for emerging themes.
Individual Adoption: Individual healthcare providers take clinically appropriate action. | Up to 6 months across implementation.
  Proportion of response by healthcare providers to the RELIEF alerts.
Appropriateness: RELIEF is seen to fit, be relevant for, or be compatible across a wide variety of settings in Canada. | Up to 6 months across implementation.
  CFIR interviews.
Fidelity. | Immediately after the intervention.
  RELIEF was implemented as intended, measured by whether the patients had their symptoms addressed by a healthcare provider.
Penetration. | Immediately after the intervention.
  Proportion of patients recruited to join RELIEF and proportion of healthcare providers participating in RELIEF at each of the sites will be assessed.
Sustainability: RELIEF is seen to be sustainable post-study. | Immediately after the intervention.
  CFIR interviews will be used.

SECONDARY OUTCOMES:
Active Participation: patients become active participants in their health monitoring and self-care through regular remote self-reporting of symptoms via RELIEF. | Up to 6 months across implementation.
  How many time patients used the RELIEF App.
Distress: Patients and their families experience less worry and concern knowing that their symptoms are being followed up by their clinical team and have access to professional opinions and treatment by their team. | Up to 6 months across implementation.
  A linear mixed model will be used to assess repeating distress scores.
Patient preferences will be measured through the Medical Maximizer-Minimizer Scale (MMS). | Immediately after the intervention.
  This scale assesses patient preferences for active vs. passive approaches to healthcare and predicts healthcare. It consists of 10 statements and identified 3 patient groups - minimizers, moderate maximizers and strong maximizers. Medical maximizers (people scoring highly on the MMS) prefer to receive more health care visits, medications, tests, and treatments, whereas minimizers prefer fewer services.
Guided Transitions: Patients avoid unnecessary trips to the emergency department for acute symptom burden through the clinical intervention made possible by RELIEF. | Up to 6 months across implementation.
  Measured via comparing the ratio of unnecessary to actual number of emergency department visits during the intervention period compared to a matched cohort.
  Unnecessary preventable visits were defined as: (1) Conditions for which exacerbations that result in hospital use suggest lack of access to adequate primary care, (2) Low-acuity visits, triaged as non-urgent at ED registration.
Satisfaction: Patients and healthcare providers are satisfied with using RELIEF for remote symptom monitoring. | 2 months following implementation and immediately afterward.
  Two month check-in and debrief surveys (2 months into the study and at the end of the study).
High Patient Engagement: Patients are engaged with RELIEF. | Up to 6 months across implementation.
  Engagement will be measured by the time patients spend on their scheduled self-assessments, or lack of time spent.
Navigation: Patients experience more seamless navigation through the healthcare system as RELIEF allows them to easily remotely self-report their symptoms and receive clinical intervention if appropriate. | 2 months following end of data collection.
  End of study surveys will be employed.
Connectedness to healthcare team. Patients feel a sense of connection with their healthcare team, which will provide comfort in knowing the team is there for them. | 2 months following implementation and immediately after data collection.
  Check in and debrief (at the end of the study) surveys will be used.
Improved palliative patient management. | Up to 6 months across implementation.
  Time between 1st email indicating alert, and 2nd email indicating alert was acknowledged (how quickly alerts were responded by healthcare providers).
Increase healthcare system capacity - RELIEF allows a single healthcare provider to oversee and follow up with a greater number of patients by improved allocation of health care resources. | Immediately after the intervention.
  Number of patients that are being followed up by a single healthcare provider.
Reduced tertiary healthcare utilization and increased healthcare cost avoidance as a result of using RELIEF. | Up to 6 months across implementation.
  Number of visits to the emergency department and associated costs, compared to matched cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Chasen, MBChB, MPhil, Principal Investigator — William Osler Health System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanuseputro P, Beach S, Chalifoux M, Wodchis WP, Hsu AT, Seow H, Manuel DG. Associations between physician home visits for the dying and place of death: A population-based retrospective cohort study. PLoS One. 2018 Feb 15;13(2):e0191322. doi: 10.1371/journal.pone.0191322. eCollection 2018. PMID 29447291
- [Background] Mooney K, Berry DL, Whisenant M, Sjoberg D. Improving Cancer Care Through the Patient Experience: How to Use Patient-Reported Outcomes in Clinical Practice. Am Soc Clin Oncol Educ Book. 2017;37:695-704. doi: 10.1200/EDBK_175418. PMID 28561689
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Tanuseputro P, Wodchis WP, Fowler R, Walker P, Bai YQ, Bronskill SE, Manuel D. The health care cost of dying: a population-based retrospective cohort study of the last year of life in Ontario, Canada. PLoS One. 2015 Mar 26;10(3):e0121759. doi: 10.1371/journal.pone.0121759. eCollection 2015. PMID 25811195
- [Background] Walker H, Anderson M, Farahati F, Howell D, Librach SL, Husain A, Sussman J, Viola R, Sutradhar R, Barbera L. Resource use and costs of end-of-Life/palliative care: Ontario adult cancer patients dying during 2002 and 2003. J Palliat Care. 2011 Summer;27(2):79-88. PMID 21805942
- [Background] Bhargava R, Keating B, Isenberg SR, Subramaniam S, Wegier P, Chasen M. RELIEF: A Digital Health Tool for the Remote Self-Reporting of Symptoms in Patients with Cancer to Address Palliative Care Needs and Minimize Emergency Department Visits. Curr Oncol. 2021 Oct 21;28(6):4273-4280. doi: 10.3390/curroncol28060363. PMID 34898539
- [Background] Isenberg SR, Tanuseputro P, Spruin S, Seow H, Goldman R, Thavorn K, Hsu AT. Cost-effectiveness of Investment in End-of-Life Home Care to Enable Death in Community Settings. Med Care. 2020 Aug;58(8):665-673. doi: 10.1097/MLR.0000000000001320. PMID 32520768
- [Background] Isenberg SR, Meaney C, May P, Tanuseputro P, Quinn K, Qureshi D, Saunders S, Webber C, Seow H, Downar J, Smith TJ, Husain A, Lawlor PG, Fowler R, Lachance J, McGrail K, Hsu AT. The association between varying levels of palliative care involvement on costs during terminal hospitalizations in Canada from 2012 to 2015. BMC Health Serv Res. 2021 Apr 13;21(1):331. doi: 10.1186/s12913-021-06335-1. PMID 33849539
- [Background] Isenberg SR, Lu C, McQuade J, Chan KKW, Gill N, Cardamone M, Torto D, Langbaum T, Razzak R, Smith TJ. Impact of a New Palliative Care Program on Health System Finances: An Analysis of the Palliative Care Program Inpatient Unit and Consultations at Johns Hopkins Medical Institutions. J Oncol Pract. 2017 May;13(5):e421-e430. doi: 10.1200/JOP.2016.014860. Epub 2017 Feb 28. PMID 28245147
- [Background] Ownby KK. Use of the Distress Thermometer in Clinical Practice. J Adv Pract Oncol. 2019 Mar;10(2):175-179. Epub 2019 Mar 1. PMID 31538028
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Anderson F, Downing GM, Hill J, Casorso L, Lerch N. Palliative performance scale (PPS): a new tool. J Palliat Care. 1996 Spring;12(1):5-11. PMID 8857241
- [Background] Jang RW, Caraiscos VB, Swami N, Banerjee S, Mak E, Kaya E, Rodin G, Bryson J, Ridley JZ, Le LW, Zimmermann C. Simple prognostic model for patients with advanced cancer based on performance status. J Oncol Pract. 2014 Sep;10(5):e335-41. doi: 10.1200/JOP.2014.001457. Epub 2014 Aug 12. PMID 25118208
- [Background] Meyers DC, Durlak JA, Wandersman A. The quality implementation framework: a synthesis of critical steps in the implementation process. Am J Community Psychol. 2012 Dec;50(3-4):462-80. doi: 10.1007/s10464-012-9522-x. PMID 22644083
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Philip J, Smith WB, Craft P, Lickiss N. Concurrent validity of the modified Edmonton Symptom Assessment System with the Rotterdam Symptom Checklist and the Brief Pain Inventory. Support Care Cancer. 1998 Nov;6(6):539-41. doi: 10.1007/s005200050212. PMID 9833305
- [Background] Donovan KA, Grassi L, McGinty HL, Jacobsen PB. Validation of the distress thermometer worldwide: state of the science. Psychooncology. 2014 Mar;23(3):241-50. doi: 10.1002/pon.3430. Epub 2013 Nov 11. PMID 25160838
- [Background] Chambers SK, Zajdlewicz L, Youlden DR, Holland JC, Dunn J. The validity of the distress thermometer in prostate cancer populations. Psychooncology. 2014 Feb;23(2):195-203. doi: 10.1002/pon.3391. Epub 2013 Sep 12. PMID 24027194
- [Background] Tittle MB, McMillan SC, Hagan S. Validating the brief pain inventory for use with surgical patients with cancer. Oncol Nurs Forum. 2003 Mar-Apr;30(2):325-30. doi: 10.1188/03.ONF.325-330. PMID 12692666
- [Background] Chen YW, HajGhanbari B, Road JD, Coxson HO, Camp PG, Reid WD. Reliability and validity of the Brief Pain Inventory in individuals with chronic obstructive pulmonary disease. Eur J Pain. 2018 Nov;22(10):1718-1726. doi: 10.1002/ejp.1258. Epub 2018 Jun 22. PMID 29883526
- [Background] Pelayo-Alvarez M, Perez-Hoyos S, Agra-Varela Y. Reliability and concurrent validity of the Palliative Outcome Scale, the Rotterdam Symptom Checklist, and the Brief Pain Inventory. J Palliat Med. 2013 Aug;16(8):867-74. doi: 10.1089/jpm.2012.0625. Epub 2013 Jun 28. PMID 23808642
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Birken SA, Powell BJ, Presseau J, Kirk MA, Lorencatto F, Gould NJ, Shea CM, Weiner BJ, Francis JJ, Yu Y, Haines E, Damschroder LJ. Combined use of the Consolidated Framework for Implementation Research (CFIR) and the Theoretical Domains Framework (TDF): a systematic review. Implement Sci. 2017 Jan 5;12(1):2. doi: 10.1186/s13012-016-0534-z. PMID 28057049
- [Background] Gruneir A, Bell CM, Bronskill SE, Schull M, Anderson GM, Rochon PA. Frequency and pattern of emergency department visits by long-term care residents--a population-based study. J Am Geriatr Soc. 2010 Mar;58(3):510-7. doi: 10.1111/j.1532-5415.2010.02736.x. PMID 20398120
- See also: Cancer Care Ontario Symptom Assessment Tools — https://www.cancercareontario.ca/en/guidelines-advice/symptom-side-effect-management/symptom-assessment-tool
- See also: Questions & Answers (Q&A), Instructions & Definitions for Use of Palliative Performance Scale — https://victoriahospice.org/wp-content/uploads/2020/08/PPSv2-QA-Instructions-and-Definitions-updated-July-2020.pdf
- See also: The Golds Standard Framework — https://www.goldstandardsframework.org.uk/cd-content/uploads/files/General%20Files/Prognostic%20Indicator%20Guidance%20October%202011.pdf
- See also: Phase 1 site assessments will be informed by the Hexagon Tool, a framework that assesses the fit and feasibility for organizations to implement an intervention — http://qic-ag.org/wp-content/uploads/2017/05/NIRN-TheHexagonTool_0.pdf
- See also: Platform where online surveys will be completed — https://www.qualtrics.com/
- See also: Phase 3 CFIR interviews informed by these guidelines — https://cfirguide.org/